CLINICAL TRIAL: NCT02808572
Title: New Biomarkers of Bone and Mineral Metabolism as Risk Factors for Morbidity/Mortality in Chronic Kidney Disease Patients Not Requiring Dialysis
Brief Title: New Biomarkers of Bone Mineral Metabolism as Cardiovascular Risk Factors in Chronic Kidney Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UF9125
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; vascular calcifications; cardiovascular risk
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vascular Calcification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular risk evaluation (Experimental): Measurement at inclusion of plasma osteoprotegerin level, plasma fibroblast growth factor 23 level, vascular calcification score and record of cardiovascular events during the 3 year follow-up
  Interventions: Biological: Plasma osteoprotegerin level; Biological: Plasma fibroblast growth factor 23 level; Procedure: Vascular calcification score

INTERVENTIONS:
Biological: Plasma osteoprotegerin level — dosage of plasma osteoprotegerin
Biological: Plasma fibroblast growth factor 23 level — dosage of plasma fibroblast growth factor 23
Procedure: Vascular calcification score — measurement of vascular calcification score by multidetection computerized tomography

SUMMARY:
To evaluate the relationships between bone mineral metabolism markers (osteoprotegerin, fibroblast growth factor 23) at inclusion and the occurence of cardiovascular events during a 7 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has signed the written consent form
* Patient with chronic renal failure defined by glomerular filtration rate (GFR) but without dialysis therapy

Exclusion Criteria:

* Pregnancy
* Patient with chronic renal failure requiring dialysis therapy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-03-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Occurence of at least one cardiovascular event during the 7 year follow-up according to osteoprotegerin level at inclusion | 7 years after inclusion
  osteoprotegerin will be measured in picomol/L

SECONDARY OUTCOMES:
Occurence of at least one cardiovascular event during the 7 year follow-up according to fibroblast growth factor 23 level at inclusion | 7 years after inclusion
  fibroblast growth factor 23 will be measured in RU/milliliter
Occurence of at least one cardiovascular event during the 7 year follow-up according to vascular calcification score at inclusion | 7 years after inclusion
Mortality | 7 years after inclusion
Kidney functions | during the 7 year follow-up
  values of creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Principal Investigator — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE
Locations (7):
- France (7):
  - AIDER, Montpellier
  - CHU Montpellier, Cardiology department, Montpellier
  - CHU Montpellier, Endocrinology department, Montpellier
  - CHU Montpellier, Intensive care unit, Montpellier
  - CHU Montpellier, Internal medicine department, Montpellier
  - CHU Montpellier, Nephrology department, Montpellier
  - AIDER, Saint-Jean-de-Védas

IPD SHARING:
Plan to Share IPD: No